CLINICAL TRIAL: NCT03182608
Title: Ultrasound Assessment of the Anatomic Landmarks for Spinal Anesthesia in Patients With Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, associate professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 16-2017-46
Record Dates: First submitted 2017-05-26; First posted 2017-06-09 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Crossover
Who Masked: Participant, Outcomes Assessor
Masking Description: An investigator evaluate the interspinous level using anatomic landmarks, then other independent investigator assess the consistency of the landmarks-guided interspinous level with the actual one using ultrasonography. Participants are blinded to the assessment results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): In the lateral decubitus position, an investigator evaluate the L4-5 interspinous level using an anatomic landmark (Tuffier's line), and then evaluate the L4-5 interspinous level using another anatomic landmark (Tenth rib line). Another investigator evaluate the actual L4-5 interspinous level by noninvasive ultrasonography.
  Interventions: Diagnostic Test: Noninvasive ultrasound assessment
- Group 2 (Experimental): In the lateral decubitus position, an investigator evaluate the L4-5 interspinous level using an anatomic landmark (Tenth rib line), and then evaluate the L4-5 interspinous level using another anatomic landmark (Tuffier's line). Another investigator evaluate the actual L4-5 interspinous level by noninvasive ultrasonography.
  Interventions: Diagnostic Test: Noninvasive ultrasound assessment

INTERVENTIONS:
Diagnostic Test: Noninvasive ultrasound assessment — An investigator evaluate the L4-5 interspinous level using anatomic landmarks in turn, then another independent investigator assess the consistency of the landmarks-guided interspinous level with the actual one by noninvasive ultrasound assessment.

SUMMARY:
Investigators assess the anatomic landmarks for spinal anesthesia in patients with hip fracture using ultrasonography.

DETAILED DESCRIPTION:
Investigators evaluate the anatomic landmarks using Tuffier's line and the tenth rib line for spinal anesthesia in patients with hip fracture, and then assess the consistency of the landmarks-guided interspinous levels with the actual interspinous level using ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for hip fracture surgery under spinal anesthesia

Exclusion Criteria:

* Anatomic abnormalities or masses in the spine
* History of spinal surgery of compression fracture

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of each anatomic landmark (Tuffier's line and tenth rib line). | Baseline
  Actual interspinous levels of the landmark-guided approches (Tuffier's line and tenth rib line) are assessed using ultrasonography.

SECONDARY OUTCOMES:
The estimation ratio related to the intervertebral levels | Baseline
  Actual interspinous levels of the landmark-guided approches (Tuffier's line and tenth rib line) are assessed using ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Hwang, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No